CLINICAL TRIAL: NCT03708263
Title: A Single-blinded, Monocentric, Randomized Pilot Study, to Evaluate the Yellow Laser PHOTOLASE PLV-585nm Versus the Reference Green Laser (KTP Excel V 532 nm) in the Treatment of Erythematotelangiectatic Rosacea
Brief Title: Evaluation of the New Laser PHOTOLASE PLV-585nm for the Treatment of Rosacea
Acronym: ROSAPHOTOLASE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: departure of Pr MORDON from the ONCOTHAI unit
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Medical Research Fund of the Tampere University Hospital, Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017_57; 2018-A01904-51 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Erythematotelangiectatic Rosacea
Keywords: 532 nm green Laser; 585 nm yellow laser; rosacea; telangiectasis score; skin disease
MeSH Terms: conditions — Rosacea; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 532nm KTP Laser (Active Comparator): Cutera® Excel V 532 nm Application of light spots 5 to 7 mm for a pulse duration of 8 to 20 ms and a fluence of 7.4 to 10 J / cm2.
  Interventions: Device: Excel V 532nm (KTP) green Laser
- 585 nm yellow laser (Experimental): PHOTOLASE PLV 585 nm Application of light spots 1.4mm for a pulse duration of 10 to 100 ms and a fluence of 0 to 65 J / cm2.
  Interventions: Device: PHOTOLASE PLV 585 nm yellow laser

INTERVENTIONS:
Device: Excel V 532nm (KTP) green Laser — Each subject's face will be divided in half and labeled as A (Right Side of the Face) or B (Left Side of Face). The allocation of active comparator and experimental treatment arms will be determined by randomization
  Arms: 532nm KTP Laser
Device: PHOTOLASE PLV 585 nm yellow laser — Each subject's face will be divided in half and labeled as A (Right Side of the Face) or B (Left Side of Face). The allocation of active comparator and experimental treatment arms will be determined by randomization
  Arms: 585 nm yellow laser

SUMMARY:
Rosacea is a frequent dermatological condition, with a chronic and disturbing evolution that is characterized by redness, permanent erythema associated with telangiectasia (visible and permanent dilatation of the small vessels). It frequently affects men and women with fair skin and can have significant psycho-emotional consequences.

To counteract the unaesthetic appearance of redness and eliminate telangiectasia, the use of the laser is proposed to the patient.

This study is a single center prospective, randomized, controlled split face study to compare 532nm KTP laser versus 585 nm PLV Laser in terms of improvement of the symptoms in the treatment of Erythematotelangiectatic Rosacea 20 subjects will receive up to 3 laser treatments at day 0, month 2 and 4 and will be followed at month 6 and 12.

DETAILED DESCRIPTION:
Adult male and female subjects 18 years of age or older will participate in the study after the objectives, methods, and potential risks of the study have been explained, and after they have signed the informed consent form.

Patients will come to the investigation center for a maximum of 6 visits.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I - III
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrolment and during the entire course of the study.
* Clinical diagnosis of Erythematotelangiectatic Rosacea stade II
* Homogeneous extend and staining telangiectasia in each half face
* Patient never treated with laser for Rosacea
* Patient doesn't wish to use systemic corticosteroids or retinoids; or topical corticosteroids or retinoids on the treated area.
* Patient agreeing to have limited exposure to the sun and use of a protective screen (index 50 or higher) every day of the study and throughout its duration if it takes place from May to September.
* Patient must be able to read, understand and sign the Informed Consent Form
* Patient able to adhere to the program of visits of the study and the other imperatives of the protocol
* Patient accepting to have photographs taken on the face
* Quality of social insurance or social security entitlement

Exclusion Criteria:

* Pregnant and/or breastfeeding woman or childbearing age without effective contraception
* Alcohol abuse assessed at the discretion of the investigator
* History of prior laser or light based procedures for any other pathology for the face within 6 months of study participation Fitzpatrick Type IV à VI
* Systemic use of isotretinoin in the 6 months prior to inclusion in the study.
* Topical use of retinoids and / or corticosteroids in the 4 weeks prior to inclusion in the study.
* Patient under photo sensitization treatment
* Patient suffering from significant concurrent illness such as type 1 diabetes, cardiovascular disease, uncontrolled hypertension, neurological disease, lupus erythematosus, scleroderma.
* Patient subject to hypertrophic or abnormal scarring
* Patient presenting or having a malignant tumor or skin cancer in the area to be treated.
* Having a known anticoagulative condition or taking prescription anticoagulation medications.
* Participation to another clinical study involving a laser or drug within three months of inclusion in the study.
* Smoker or former smoker in the 12 months prior to inclusion in the study.
* Patient with excessive tattoos in the area to be treated and / or wishing to tattoo the treated area during the study.
* Patient treated for cancer by chemotherapy or radiotherapy
* Patient with hyper or hypo pigmentation
* Patient unable to understand protocol or give consent
* Legal incapacity (persons deprived of their liberty or under guardianship or curatorship)
* Patient in emergency or in detention
* Clinical follow-up impossible for psychological, family matters, social or geographical reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Degree of improvement in Erythematotelangiectatic Rosacea | at Month 2
  Measured, for each treatment arm, based on blinded physician assessment of subject photographs using the 7 points Telangiectasia Grading Score.
  (-1 = Aggravation of telangiectasia, 0 = no change, 1 = poor improvement (<25% decrease), 2 = intermediate improvement (25-50% decrease), 3 significant improvement (50-75% decrease), 4 = very significant improvement (75-99% decrease), 5 = complete improvement (100% decrease)

SECONDARY OUTCOMES:
Degree of improvement in Erythematotelangiectatic Rosacea evaluated by a blinded physician. | at Month 4, 6,12
  Measured, for each treatment arm, based on subject photographs using the 7 points Telangiectasia Grading Score
Measures of skin reaction for each treatment arm | At baseline, At Month 2, At Month 4 (if realized)
  Measured with a 4 points scale : no reaction, low, moderate and severe reaction
Pain evaluation during each treatment | At baseline, At Month 2, At Month 4 (if realized)
  Mosby Pain Rating Scale for each treatment arm
Change in lesion skin color in each treatment arm | At Baseline, at Month 2, 4, 6,12
  Measured with Chroma-Meter CR400 (Konica Minolta), Mean a* value
Subject satisfaction level | At Month 6,12
  Comparison of each treatment arm using Subject Overall Evolution Scale
Change in Life Quality | At Selection, at Baseline, at Month 2, 4 (if realized), 6,12
  Comparison of Dermatology Life Quality Index
Practitioner's opinion | At baseline, At Month 2, At Month 4 (if realized)
  Comparison, for each treatment arm, of comfort of use, practicality, duration of treatment
Adverse Events | At Baseline, At Month 2, 4, 6,12
  Incidence and severity of adverse effects, for each treatment arm, during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Cyril MAIRE, MD, Principal Investigator — University Hospital, Lille; Serge MORDON, Pr, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France